CLINICAL TRIAL: NCT00317759
Title: Phase I Study to Evaluate the Safety of Cellular Adoptive Immunotherapy Using Autologous CD8+ Antigen-Specific T Cell Clones Following Fludarabine Lymphodepletion for Patients With Metastatic Melanoma
Brief Title: Fludarabine Followed By Adoptive Immunotherapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1796.00; FHCRC-1796.00; CDR0000327817 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2010-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — fludarabine phosphate

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Biological therapies such as cellular adoptive immunotherapy use different ways to stimulate the immune system and stop cancer cells from growing. Fludarabine may help the immune system kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of fludarabine followed by cellular adoptive immunotherapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and toxicity of adoptive immunotherapy comprising autologous CD8+ antigen-specific cytotoxic T-lymphocyte (CTL) clones after fludarabine in patients with stage IV melanoma.
* Determine the duration of in vivo persistence of these CTL clones in these patients.

Secondary

* Determine the antitumor effect of this regimen in these patients.

OUTLINE: This is an open-label, nonrandomized study.

Patients undergo leukapheresis or weekly phlebotomy for the collection of peripheral blood mononuclear cells from which autologous antigen-specific CD8+ cytotoxic T-lymphocyte (CTL) clones are generated. Patients receive autologous antigen-specific CD8+ CTL clones IV over 30-60 minutes on days 0 and 21 in the absence of rapid disease progression or unacceptable toxicity. Patients also receive fludarabine IV once daily on days 14-18.

Patients are followed for up to 1 year.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma

  * Stage IV disease
* HLA-A2 or -A3-expressing disease
* Bidimensionally measurable residual disease by palpation or radiographic imaging (e.g., x-ray or CT scan)
* No CNS metastases

  * Previously treated CNS involvement allowed provided there is no evidence of CNS disease at least 2 months after completion of therapy

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* Karnofsky 80-100%

Life expectancy

* More than 6 months

Hematopoietic

* Platelet count > 100,000/mm^3
* Absolute neutrophil count > 2,000/mm^3

Hepatic

* SGOT no greater than 3 times upper limit of normal
* Bilirubin no greater than 1.6 mg/dL
* INR no greater than 1.5 times normal

Renal

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No congestive heart failure
* No clinically significant hypotension
* No symptoms of coronary artery disease
* No cardiac arrhythmia by EKG requiring drug therapy

Pulmonary

* No clinically significant pulmonary dysfunction
* FEV_1 at least 1.0 L*
* DLCO at least 45%* NOTE: *For patients with a history of pulmonary dysfunction

Immunologic

* No active infection
* No oral temperature greater than 38.2°C within the past 48 hours
* No systemic infection requiring chronic maintenance or suppressive therapy

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy (e.g., interleukins, interferons, melanoma vaccines, IV immunoglobulins, expanded polyclonal tumor-infiltrating lymphocytes, or lymphokine-activated killer therapy)

Chemotherapy

* At least 3 weeks since prior chemotherapy (standard or experimental)

Endocrine therapy

* No concurrent steroids

Radiotherapy

* At least 3 weeks since prior radiotherapy

Surgery

* Not specified

Other

* At least 3 weeks since prior immunosuppressive therapy
* No concurrent pentoxifylline
* No other concurrent investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2003-05; Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Wallen H, Thompson JA, Reilly JZ, Rodmyre RM, Cao J, Yee C. Fludarabine modulates immune response and extends in vivo survival of adoptively transferred CD8 T cells in patients with metastatic melanoma. PLoS One. 2009;4(3):e4749. doi: 10.1371/journal.pone.0004749. Epub 2009 Mar 9. PMID 19270751